CLINICAL TRIAL: NCT02274415
Title: Study of the Immunogenicity of a Prime Boost Vaccination Strategy Combining Conjugated Anti-pneumococcal and Polysaccharide Anti-pneumococcal Vaccine Compared to Polysaccharide Anti -Pneumococcal Vaccine Alone in Patients With Sickle Cells Disease
Brief Title: Immunogenicity Study of an Anti-pneumococcal Vaccination Strategy in Patients With Sickle Cells Disease
Acronym: DREVAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AOM10028; P100105 (Other: Assistance Publique Hôpitaux de Paris)
Record Dates: First submitted 2014-09-22; First posted 2014-10-24 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2017-10

CONDITIONS: Invasive Pneumococcal Infections; Sickle Cells Disease
Keywords: Streptococcus pneumoniae; Sickle cell disease; Immunogenicity; Antibody response
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Vaccination; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCV vaccine following by the PSV vaccine (Experimental): Group 1: patients will receive a first boost with 13-valent pneumococcal conjugate vaccine (PCV) (one dose at W0) and then one administration of the PSV vaccines (one dose at W4).
  Interventions: Biological: Vaccination with the combined vaccine (Prevenar13 ®); Biological: Vaccination with the polysaccharide vaccine (Pneumo 23 ®)
- vaccine Pneumo 23 (Active Comparator): Group 2: patients will receive a single administration of 23-valent pneumococcal polysaccharide vaccine (PSV) (one dose at W4)
  Interventions: Biological: Vaccination with the polysaccharide vaccine (Pneumo 23 ®)

INTERVENTIONS:
Biological: Vaccination with the combined vaccine (Prevenar13 ®)
  Arms: PCV vaccine following by the PSV vaccine
Biological: Vaccination with the polysaccharide vaccine (Pneumo 23 ®)

SUMMARY:
Streptococcus pneumoniae is the major cause of bacterial infection in patients with sickle cells disease.

The 23-valent pneumococcal polysaccharide vaccine (PSV) is supposed to be poorly immunogenic in these patients. We want to evaluate whether a prime with a 13-valent pneumococcal conjugate vaccine (PCV), able to induce immunologic memory, would improve the immune response against SP polysaccharides (SPP).

Primary objective: To evaluate and compare the specific antibody response to a prime-boost vaccine strategy combining PCV prime at W0 followed by the administration of PSV boost at W4, to the administration of PSV alone at W4 in patients with sickle cells disease.

Secondary objectives: Evaluation and comparison of the specific antibody response to the thirteen pneumococcal serotypes shared by the PCV and PSV vaccines, 4 weeks after the single PSV vaccination for patients from Group 1 or 4 weeks after the boost PSV vaccination for patients from group 2. Evaluation of the duration of the specific antibody response at W24 and 96. Evaluation of the T CD4 lymphocyte response to the CRM 197 protein. Safety of the vaccines.

Study Design: Randomised, monocentric, controlled phase II study of the immunological efficacy of a prime boost strategy combining the sequential administration of the PCV and PSV, compared to the administration of the PSV alone. 180 adults patients with sickle cells disease will be included. The primary endpoint : proportion of responders at W8 to at least 10 of thirteen serotypes. Secondary endpoints : Proportion of responders at W8 according to 4 categories of responders: 5-7; 3-4; 2-1 and 0. Evaluation of the pneumococcal opsonophagocytic activity (OPA) at baseline and W8 for each serotype, defined as the proportion of patients with OPA > 1:8 geometric mean of the specific antibody titers proportion of patients who experienced an increase of specific antibody levels 1 g/ml. Evaluation of the priming effect of the PCV vaccine in the group 1. Duration of the specific antibody responses at week 24 and W96. CD4 T lymphocyte responses to the CRM 197 protein (proliferative and cytokine production) at weeks 0, 8 and 12. Safety of the vaccines frequency of Streptococcus pneumoniae infections.

Statistical Considerations: With a sample size of 180 patients, and a randomization ration of 1:1, the study will have a power of at least 90% to show a difference of 25% category between the group receiving PCV and PSV vs the group receiving PSV alone (two-sided type I error = 5%). The primary comparison between both groups will be performed using a Chi2 test for independent groups or a Fisher exact test where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Adult patient with sickle cell anemia (SS homozygous, SC heterozygous compound Sbetathal heterozygous)

Exclusion Criteria:

* Heterozygous sickle cell anemia
* Active infection
* Hypersensitivity known or suspected to Prevenar 13® or to Pneumo 23® or to any of the excipients included in the formulation or in the administration system
* Coagulation abnormality indicating against an intramuscular injection (Platelets <50 000 or TP<50%)
* Current chemotherapy or radiotherapy, except for using Siklos®/Hydrea® in the context of sickle cell anemia
* Vaccination whatever in the last 2 months before the protocol vaccination, except influenza vaccination (within 30 days)
* Vaccination whatever, provided in the first 2 months following the protocol vaccinations, except influenza vaccination (within the first month following the protocol vaccinations))
* History of pneumococcal vaccination with Pneumo 23® in the previous year
* End-stage renal failure(dialyzed patient, clearance<10ml/mn)
* HIV infection at baseline
* Pregnancy or breastfeeding (A dosage of betaHCG will be conducted for women in childbearing age),contraception recommendation the first 8 weeks of the test for women in childbearing age
* Participation in a clinical research protocol using a drug within the month prior to inclusion.
* No medical assurance
* Adults under tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
the proportion of responders at least to 10 of thirteen serotypes | at Week 8
  A responder is defined by a rise least two fold from baseline) of antibody titers specific to pneumococcal serotypes;

SECONDARY OUTCOMES:
Proportion of responders according to 4 categories of responders: 5-7; 3-4; 2-1 and 0. | at Week 8
  Response is defined as fold rise of antibody titers (W8 to baseline)
Evaluation of the pneumococcal opsonophagocytic activity (OPA) for each serotype, | at baseline and Week 8
  defined as the proportion of patients with OPA > 1:8.
The antibody response of the conjugate vaccine | at week 4
  The antibody response to the 13 serotypes of the conjugate vaccine in terms of geometric mean of the specific antibody titers (µg/ml)
The antibody response to the 13 serotypes of the conjugate vaccine in terms of proportion of patients | at week 4
In the group 1 antibodies titers (µg/ml) | at week 24 and W96
Number of T CD4 cells responsive to the CRM 197 protein (proliferative and cytokine production) in the two groups of the study | at weeks 0, 8 and 12.
Number of Streptococcus pneumoniae infections | between baseline and W96
  Number of Streptococcus pneumoniae infections (bacteremia, meningitis, pneumonia, sinusitis, upper respiratory tract infections)

CONTACTS AND LOCATIONS:
Overall Officials: Yves LEVY, PHD, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Melica G, Bartolucci P, Audureau E, Le Corvoisier P, Habibi A, Gellen J, Selmane D, Michel M, Lacabaratz C, Levy Y. Immunological Efficacy of Pneumococcal Vaccination Including the 13-Valent Pneumococcal Conjugate Vaccine in Adult Patients With Sickle Cell Disease: Results of the Randomized DREVAC Controlled Trial. Clin Infect Dis. 2023 Jun 8;76(11):1949-1958. doi: 10.1093/cid/ciad037. PMID 36705266